CLINICAL TRIAL: NCT06191302
Title: Investigation of COVID-19 Post-acute Sequelae in Patients From Hvidovre Hospitals Catchment Area, and in a Register of the Danish Population 2000-2026
Brief Title: Post-acute COVID-19 Sequelae in Denmark
Status: Recruiting | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Ove Andersen, Research Director, professor,, Hvidovre University Hospital
Other Study IDs: H-24039578
Record Dates: First submitted 2024-01-02; First posted 2024-01-05 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Non-communicable Disease; COVID-19
Keywords: Sequelae; Inflammation; Ageing; Non-communicable disease
MeSH Terms: conditions — Noncommunicable Diseases; COVID-19; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SARS-CoV-2 positive patients: a cohort of former patients hospitalized with COVID-19
  Interventions: Procedure: blood sample; Other: Online questionaire
- SARS-CoV-2 negative patients: a control group of former patients hospitalized with other respiratory diseases
  Interventions: Procedure: blood sample; Other: Online questionaire

INTERVENTIONS:
Procedure: blood sample — Blood sample collected in the post-acute period (follow-up visit) will be analysed for biomarkers predictive for diseases related to and disease progression in various organ systems (e.g., cardiovascular, pulmonary, and renal systems), including e.g., Pro-BNP, NGAL, and interleukins.
Other: Online questionaire — The participants will complete an online questionnaire related to disease and health issues associated with COVID-19 and COVID-19 post-acute sequalae's and existing Non-Communicable Disease.

SUMMARY:
Since the first SARS-CoV-2 cases in 2019, over 660 million COVID-19 cases have been reported globally, including 183 million in the EU. Up to 70% of those infected experience reduced organ function four months or more after a COVID-19 diagnosis, potentially increasing the risk of non-communicable diseases (NCDs). The post-acute phase (PAP) after COVID-19 (four months or more after the acute phase) can lead to impaired function in various organ systems, with a focus on the lungs, cardiovascular system, and kidneys. These three NCDs collectively impose a significant burden on individuals and society. Urgently, we need to understand the connection between COVID-19, PAP and NCDs, identifying robust biomarkers for early detection. This study examines PAP and associated risk factors, investigating the link between PAP and the heightened risk of lung, heart, and kidney complications. Utilizing data from a cohort of COVID-19 patients and a control group with respiratory diseases, the study aims to determine prevalence and risk ratios more precisely. The aim is to contribute to minimizing the risk of NCD development or exacerbation in current and future COVID-19 patients, enhancing our understanding of chronic disease development at the population leve

DETAILED DESCRIPTION:
The post-acute phase (PAP) after COVID-19 (four months or more after the acute phase of COVID-19) can manifest with reduced function in multiple organ systems, with a particular focus on the lungs, cardiovascular system, and kidneys. Collectively, these three non-communicable diseases (NCDs) represent a significant burden for both the individual and society as a whole. There is an urgent need to elucidate this connection and build a more detailed understanding of the link between COVID-19's PAP and individual NCDs, as well as to identify robust biomarkers that can assist in the early identification of the development of these NCDs.

This study focuses on PAP and the associated risk factors in this later phase of the disease, examining the relationship between PAP and the increased risk of specifically lung, heart, and kidney complications in the Danish population. Additionally, data (medical records, registry data, patient reported outcomes and blood samples) from a cohort of former patients hospitalized with COVID-19, as well as a control group hospitalized with other respiratory diseases, are investigated to determine the prevalence and risk ratios in disease development more precisely.

The purpose of the study is to contribute to minimizing the risk of developing or worsening NCDs in current and future COVID-19 patients, as well as contributing to our understanding of chronic disease development at the population level. The study aims to investigate the hypothesis that biomarkers can predict if SARS-CoV-2 infection leads to increased and exacerbated non-communicable pulmonary, cardiovascular, and renal diseases.

Further, we address the unmet need to understand the molecular mechanisms responsible for the link between post-acute effects of SARS-CoV-2 and complications in the pulmonary, cardiovascular, and renal system. More specific we will investigate the molecular mechanisms responsible for the aetiology and decline in organ function.

The population in the registry study is the entire population of Denmark. The population in the clinical cohort consists of former patients who have been admitted to Hvidovre Hospital with the diagnosis OBS COVID. Participants consent to the use of residual material from their blood sample, taken during their hospitalization with the diagnosis OBS-COVID in the period 2020-2022 (index blood sample). After obtaining consent, patients come to Hvidovre Hospital, where a blood sample (follow-up blood sample) is taken, and an online questionnaire is completed and stored in REDCap. Blood samples are analyzed and compared with collected registry data and questionnaire data, after which the results are reported in international peer-reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

* Has a blood sample in the clinical biobank related to the OBS-COVID index admission
* Aged above 18 years at time of index-admission

Exclusion Criteria:

* Patients without a Danish personal identification number
* Patients who do not understand or speak Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participating patients are former patients admitted to Hvidovre Hospital with the diagnosis OBS-COVID
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
1.Is there a difference in the incidence and disease progression of NCD (pulmonary, cardiovascular, and renal disease) in the PAP between SARS-CoV-2-positive patients and a control group of patients admitted with other respiratory diseases? | Follow-up from index-admission to March 1, 2026
  Primary outcomes:
  * Incidence of incipient NCD
  * Change in health-state of pre-existing NCD
2. Is there a difference in the association of admission biomarkers and incidence, severity, and disease progression of NCD in PAP, between SARS-CoV-2 positive patients and a control group of patients admitted with other respiratory diseases? | Follow-up from index-admission to March 1, 2026
  • Level in admission biomarkers associated with incipient or worsening of NCD in PAP
3. Which biomarkers are involved in development or disease progression of NCDs in PAP? | Follow-up from index-admission to March 1, 2026
  Principal outcomes:
  * Identify in vivo biomarkers in admission and follow-up blood samples associated with tissue /organ damage, and inflammation
  * Investigate in vitro molecular mechanisms in follow-up blood samples by examining cellular morphology, metabolism, stress response, fibrosis, viability, proliferation, senescence, and inflammation.

OTHER OUTCOMES:
1.Is there a difference in the incidence and disease progression of NCD (pulmonary, cardiovascular, and renal disease) in the PAP between SARS-CoV-2-positive patients and a control group of patients admitted with other respiratory diseases? | Follow-up from index-admission to March 1, 2026
  Other outcomes:
  * Incidence of incipient NCD stratified by the socioeconomic position of patients
  * Change in health-state of pre-existing NCD stratified by the socioeconomic position of patients
2. Is there a difference in the association of admission biomarkers and incidence, severity, and disease progression of NCD in PAP, between SARS-CoV-2 positive patients and a control group of patients admitted with other respiratory diseases? | Follow-up from index-admission to March 1, 2026
  • Level in admission biomarkers associated with symptoms, lower quality of life, functional impairment in PAP.

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andersen, Professor, Principal Investigator — Department of Clinical Research, Copenhagen University Hospital, Hvidovre; Jon Ambaek Durhuus, PhD, Study Chair — Department of Clinical Research, Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital, Amager and Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Only aggregated data can be available for other researchers due to Danish Data Protection Law